CLINICAL TRIAL: NCT06366425
Title: Non-invasive Screening for Chronic Liver Diseases in the General Population. A Prospective Study
Brief Title: Screening for Chronic Liver Diseases in General Population
Acronym: HEPGEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: On-call medical home (MMG) Clermont-Hérault (Unknown); Medical office Montpeyroux (Unknown); Medical office Clermont-Hérault (Unknown); Medical office Aniane (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL23_0272
Record Dates: First submitted 2024-03-22; First posted 2024-04-15 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Fibrosis, Liver
Keywords: Non-alcoholic fatty liver disease (NAFLD); Hepatocellular carcinoma (HCC); Chronic liver diseases; Linkage to care; Fibrosis research; Non-invasive diagnosis; FIB-4; Fibroscan
MeSH Terms: conditions — Liver Cirrhosis; Non-alcoholic Fatty Liver Disease; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Population with a chronic liver disease risk factor (Other): Patient aged ≥ 40 years, with no known liver disease, consulting a general practitioner and having at least one risk factor for chronic liver disease: risky consumption of alcoholic beverages according to the AUDIT questionnaire, the presence of a metabolic syndrome, diabetes or a risk factor for viral hepatitis B/D or C.
  Interventions: Diagnostic Test: Blood sample then fibroscan

INTERVENTIONS:
Diagnostic Test: Blood sample then fibroscan — The patient takes a blood test if none less than 6 months old is available, including a complete blood count (CBC) and a hepatic check. The FIB-4 score will be calculated from this blood test.
  If the result of the FIB-4 test is greater than 1.3 the person will be contacted by the SELHV (Service Expert de Lutte contre les Hépatites Virales) of the University Hospital of Montpellier in order to schedule, if she wishes, a second non-invasive screening examination of liver fibrosis by Fibroscan.

SUMMARY:
Improving the care of patients with liver diseases in primary care and will allow patients with chronic liver disease to benefit from a course appropriate care.

DETAILED DESCRIPTION:
The prevalence of chronic liver diseases continues to increase on the one hand by the increase in non-alcoholic fatty liver disease (NAFLD) which affects 25% of the general population as well as the increased incidence of hepatocellular carcinoma in recent years. Screening for liver fibrosis in the general population represents a major public health issue.

The FIB-4 score is obtained by a blood test. This score combines age, measurement of ALT/ASAT (alanine aminotransferase / aspartate-aminotransferase) and platelet count. This score is sensitive for detecting advanced fibrosis liver and allows 71% of patients to avoid a liver biopsy.

Transient elastometry (Fibroscan®) is another very effective non-invasive assessment in the diagnosis of chronic liver diseases and hepatic fibrosis. It has already been demonstrated by several studies that combining several non-invasive fibrosis tests allows to improve the precision of the result.

The investigators hypothesize that offering an additional assessment by Fibroscan for patients screened by a blood test (FIB-4 Score) as possibly having advanced liver fibrosis (Score >1.3) will raise awareness among professional practitioners and the general population with chronic liver diseases and refine screening for chronic liver diseases.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years
* Without known liver pathologies
* Having at least one risk factor for chronic liver disease: risky consumption of alcoholic beverages according to the AUDIT questionnaire, the presence of metabolic syndrome, diabetes or a risk factor for viral hepatitis B, D or C.

Exclusion Criteria:

* Fibroscan already performed in the last 12 months
* Failure to collect express oral consent
* Patient not affiliated with or not benefiting from a national health insurance scheme
* Patient protected by law
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Pregnant or breastfeeding woman

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2024-10-09 (Actual); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the liver fibrosis screening acceptability (FIB-4) | During the inclusion assessment at day 1 (Visit 0)
  percentage of patients who agreed to a FIB-4 blood test among all included patients offered screening.
Evaluation of the liver fibrosis screening acceptability (FIB-4 and Fibroscan) | During the inclusion assessment at day 1 (Visit 0) and at 1 month (visit 1)
  percentage of patients who agreed to a FIB-4 blood test FIB-4 followed by Fibroscan (if FIB-4 score>1.3) among all included patients offered screening.

SECONDARY OUTCOMES:
Prevalence of advanced liver fibrosis by elastometry pulse (Fibroscan®) with a FIB-4 score>1.3 | During the inclusion assessment at day 1 (Visit 0) and at 1 month (visit 1)
  If FIB-4 Score>1.3 a pulse elastometry (Fibroscan®) will be performed. A fibrotest measurement of ≥10 KPa (Kilopascals) or a score ≥F3 will be considered as advanced hepatic fibrosis.
Prevalence of excessive consumption of alcohol | During the inclusion assessment at day 1 (Visit 0)
  Excessive alcohol consumption will be evaluated by the AUDIT-C questionnaire (Alcohol Use Disorders Identification Test) with a score ranging from 0 (lower risk) to 12 (higher risk of misuse), a score of > or = 3 for women and > or = 4 for men indicates misuse.
Prevalence of a history or drug use | During the inclusion assessment at day 1 (Visit 0)
  Rate of participants with a history or current use of drugs among included patients.
  Answered by the patient face to face with the doctor.
The correlation between advanced liver fibrosis and risk factors for liver disease (presence of metabolic syndromes, viral hepatitis, alcool use disorders) | During the inclusion assessment at day 1 (Visit 0) and at 1 month (visit 1)
  The correlation will be evaluated by the rate of patients with risk factors for liver disease and advanced fibrosis, among all those who underwent Fibroscan.
  A fibrotest measurement of ≥10 KPa (Kilopascals) or a score ≥F3 will be considered as advanced hepatic fibrosis
  The presence of metabolic syndrom if at least 3 of the following risk factors are present : arterial hypertension (≥ 130/85 mmHg), hypertriglyceridemia (≥ 1.7 mmol/L), low HDL-cholesterol (Men< 1 mmol/L; women < 1.3 mmol/L) , android obesity (≥ 102 cm men; ≥ 88 cm women) and fasting hyperglycemia (> 100 mg/dL)
  Presence of an alcohol use disorders : AUDIT-C questionnaire with a score of ≥ 3 for women and ≥ 4 for men indicates misuse.
  Presence of diabetes in medical records.
  Presence of hepatitis by using a serology blood test (Hepatitis C Virus : HCV RNA, surface antigen of the hepatitis B virus : HBsAg, anti HBsAg, anti HBCAg, HBV DNA, HBeAg, anti HBeAg, Delta virus in case of hepatitis B positivity).
prevalence of viral hepatitis | During the inclusion assessment at day 1 (Visit 0) and at 1 month (visit 1)
  Diagnosis of hepatitis by using a rapid diagnostic orientation test (TROD) by collecting of a drop of blood from the fingertip which is placed on a plate with a reactive solution in order to establish the presence of antigens and/or with a serology blood test (( Hepatitis C Virus : HCV RNA, HCV+, surface antigen of the hepatitis B virus : HBsAg, anti HBsAg, anti HBCAg, HBV DNA, HBeAg, anti HBeAg, Delta virus in case of hepatitis B positivity).
  Prevalence of viral hepatitis among all included patients.
Description of socio-demographic characteristics of participants | During the inclusion assessment at day 1 (Visit 0)
  Description of the socio-demographic characteristics of people benefiting from an assessment of liver fibrosis by transient elastometry (Fibroscan®) as part of the study.
  Socio-demographic characteristics will be collected by a patient questionnaire (age, education, profession, income, health insurance, marital status, housing, living conditions) realised face to face with the doctor.

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena MESZAROS, MD, Study Director — University Hospital, Montpellier
Locations (1):
- CHU de Montpellier, Montpellier, France

REFERENCES:
- [Background] Friedrich-Rust M, Ong MF, Martens S, Sarrazin C, Bojunga J, Zeuzem S, Herrmann E. Performance of transient elastography for the staging of liver fibrosis: a meta-analysis. Gastroenterology. 2008 Apr;134(4):960-74. doi: 10.1053/j.gastro.2008.01.034. Epub 2008 Jan 18. PMID 18395077
- [Background] de Franchis R, Bosch J, Garcia-Tsao G, Reiberger T, Ripoll C; Baveno VII Faculty. Baveno VII - Renewing consensus in portal hypertension. J Hepatol. 2022 Apr;76(4):959-974. doi: 10.1016/j.jhep.2021.12.022. Epub 2021 Dec 30. PMID 35120736
- [Background] Gines P, Castera L, Lammert F, Graupera I, Serra-Burriel M, Allen AM, Wong VW, Hartmann P, Thiele M, Caballeria L, de Knegt RJ, Grgurevic I, Augustin S, Tsochatzis EA, Schattenberg JM, Guha IN, Martini A, Morillas RM, Garcia-Retortillo M, de Koning HJ, Fabrellas N, Pich J, Ma AT, Diaz MA, Roulot D, Newsome PN, Manns M, Kamath PS, Krag A; LiverScreen Consortium Investigators. Population screening for liver fibrosis: Toward early diagnosis and intervention for chronic liver diseases. Hepatology. 2022 Jan;75(1):219-228. doi: 10.1002/hep.32163. Epub 2021 Dec 10. PMID 34537988
- [Background] Dam-Larsen S, Franzmann M, Andersen IB, Christoffersen P, Jensen LB, Sorensen TI, Becker U, Bendtsen F. Long term prognosis of fatty liver: risk of chronic liver disease and death. Gut. 2004 May;53(5):750-5. doi: 10.1136/gut.2003.019984. PMID 15082596
- [Background] Teli MR, Day CP, Burt AD, Bennett MK, James OF. Determinants of progression to cirrhosis or fibrosis in pure alcoholic fatty liver. Lancet. 1995 Oct 14;346(8981):987-90. doi: 10.1016/s0140-6736(95)91685-7. PMID 7475591
- [Background] Marshall AD, Micallef M, Erratt A, Telenta J, Treloar C, Everingham H, Jones SC, Bath N, How-Chow D, Byrne J, Harvey P, Dunlop A, Jauncey M, Read P, Collie T, Dore GJ, Grebely J. Liver disease knowledge and acceptability of non-invasive liver fibrosis assessment among people who inject drugs in the drug and alcohol setting: The LiveRLife Study. Int J Drug Policy. 2015 Oct;26(10):984-91. doi: 10.1016/j.drugpo.2015.07.002. Epub 2015 Jul 16. PMID 26256938
- [Background] Mwamba-Kalambayi P, Etienne A, Chirpaz E, Gelu-Simeon M, Cuissard L, Deloumeaux J, et al. Étude comparative de la fréquence des hépatites B et C chez les personnes nouvellement diagnostiquées pour carcinome hépatocellulaire en France métropolitaine et dans les départements et régions d'outre-mer, 2015-2019. Bull Epidémiol Hebd. 2022;(3-4): 85-94.
- [Background] Oberti F, Cailliez E, Hubert I et al. Dépistage de la fibrose hépatique en populations générale et de médecine générale (étude DEFIH). Gastroenterol Clin Biol 2006;30:A7.
- See also: Recommandations pour le diagnostic et le suivi non-invasif des maladies chronique du foie, Association Française pour l'étude du foie. — https://afef.asso.fr/wp-content/uploads/2023/06/DNI-VERSION-FINALE-RECO-2020-V2.pdf